CLINICAL TRIAL: NCT01284283
Title: 2-Year Post-Approval Study to Investigate the STAR Ankle Under Actual Conditions of Use
Brief Title: 2-Year Post-Approval Study to Investigate the Scandinavian Total Ankle Replacement System (STAR) Ankle Under Actual Conditions of Use
Acronym: STAR 2 PAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Encore Medical, L.P. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STAR 2 Year
Record Dates: First submitted 2010-11-02; First posted 2011-01-26 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Primary Arthrosis; Post Traumatic Arthritis; Rheumatoid Arthritis; Osteoarthritis
Keywords: Arthrosis; Rheumatoid Arthrosis; Arthritic Joint; Rheumatoid Arthritis; Osteoarthritis; Total Ankle Replacement
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single (Other): Device: Scandinavian Total Ankle Replacement System (STAR Ankle)
  Interventions: Device: Scandinavian Total Ankle Replacement System (STAR Ankle)

INTERVENTIONS:
Device: Scandinavian Total Ankle Replacement System (STAR Ankle) — For total ankle replacement
  Other Names: STAR

SUMMARY:
This post-approval study is being conducted to examine the performance of the STAR Ankle under actual conditions of use.

DETAILED DESCRIPTION:
This investigation is a prospective, multi-center, single-arm study. 98 subjects are to be enrolled in this clinical investigation. Enrolled subjects will be assessed at Pre-Operative, Operative/Discharge, and at 6 Weeks, 6, 12, and 24 Months after the index procedure. Safety, efficacy, and effectiveness analyses will be performed for all follow-up points during the study.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe pain, loss of mobility and function of the ankle (Buechel-Pappas Scale)
* Primary arthrosis, post traumatic arthrosis or rheumatoid arthrosis
* At least six months of conservative treatment for severe ankle conditions, confirmed by the patient medical history, radiograph studies and medication record
* Willing and able to give informed consent

Exclusion Criteria:

* Patients who have not reached skeletal maturity
* Active or prior deep infection inthe ankle joint or adjacent bones
* Prior arthrodesis at the involved site
* History of prior mental illness or patient demonstrates that their mental capacity may interfere with their ability to follow the study protocol
* Obesity (weight greater than 250 lbs)
* History of current prior drug abuse or alcoholism
* Any physical condition precluding major surgery
* Hindfoot malpositioned by more than 35 degrees or forefoot malalignment which would preclude a plantigrade foot
* Lower extremity vascular insufficiency demonstrated by Doppler arterial pressure
* Avascular necrosis of the talus
* Inadequate skin coverage above the ankle joint
* Patients under the age of 35 who are unwilling or unable to accept the physical limitations imposed by ankle arthroplasty, including limitations on certain vigorous physical activities (e.g. basketball, football) and on manual labor
* Juvenile onset Type I diabetes
* Adult onset Type II diabetes when accompanied by neuropathic changes or a history of foot infection in either foot
* Pregnancy
* Avascular necrosis of the tibia
* Significant bone tumor of the foot or ankle
* Severe deformity that would not normally be eligible for ankle surgery
* Prior surgery and/or injury that has adversely affected the ankle bone stock
* Severe osteoporotic or osteopenic condition or other conditions that may lead to inadequate implant fixation in the bone
* Insufficient ligament support
* Motor dysfunction due to neuromuscular impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2009-11; Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint | 2 years
  The primary objective of this study is to examine the performance of the STAR™ Ankle under actual conditions of use, employing the approved instructions for use, labeling, and instrumentation. The principal endpoint consists of evaluating the safety and effectiveness of the STAR™ Ankle. Overall patient success is defined as:
  1. ≥ 40 point improvement in total Buechel-Pappas Scale score
  2. No device failures
  3. Radiographic success (no clinically significant radiographic evidence of loosening, tilting or migration > 4mm)
  4. No major complications

SECONDARY OUTCOMES:
Secondary Endpoints | 2 years
  In addition to the principal endpoint, information on the following efficacy outcomes will be assessed:
  * Total Buechel-Pappas Scale score
  * Pain Visual Analog Scale
  * Quality of Life
  * American Orthopaedic Foot & Ankle Society (AOFAS) Ankle Hindfoot Scale
  The following radiographic endpoints will be assessed by anterior/posterior and lateral radiographs by the treating surgeon and an independent radiographic reviewer:
  * Radiolucency
  * Migration

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Maartense, MD, Study Director — Stryker Nordic
Locations (9):
- United States (9):
  - The CORE Institute, Phoenix, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - Palo Alto Medical Research Foundation (Sutter Health), Palo Alto, California
  - Kaiser Permanente, San Francisco, California
  - William Beaumont Hospital, Royal Oak, Michigan
  - Reno Orthopaedic Center, Reno, Nevada
  - Kenneth Mroczek, MD-NYU, New York, New York
  - University of Pennsylvania Health Systems-PA Foot and Ankle Surgeons, Philadelphia, Pennsylvania
  - Center for Foot and Ankle Restoration, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No